CLINICAL TRIAL: NCT02740296
Title: Depression and Immune Function in Multiple Sclerosis (MS)
Acronym: DENIM
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: National Multiple Sclerosis Society (Other); Universitätsklinikum Hamburg-Eppendorf (Other); NeuroCure Clinical Research Center, Charite, Berlin (Other)
Responsible Party: Principal Investigator, Friedemann Paul, Prof. Dr., Charite University, Berlin, Germany
Other Study IDs: DENIM
Record Dates: First submitted 2016-04-12; First posted 2016-04-15 (Estimated); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Multiple Sclerosis; Depressive Disorder, Major
MeSH Terms: conditions — Multiple Sclerosis; Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Healthy controls: Healthy controls
  Interventions: Other: No intervention
- RRMS: Relapsing-Remitting Multiple Sclerosis
  Interventions: Other: No intervention
- RRMS+MDD: Relapsing-Remitting Multiple Sclerosis and Major Depressive Disorder
  Interventions: Other: No intervention
- MDD: Major Depressive Disorder
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention

SUMMARY:
Depression is one of the most common symptoms of multiple sclerosis (MS) with a life-time prevalence of major depressive disorder (MDD) of up to 50%. Depression occurs more frequently in MS than in other chronic diseases including other neurological and inflammatory disorders and may contribute to lower quality of life, cognitive problems, difficulties at work, and poorer long term health outcomes. Despite its clinical relevance, the biological mechanisms which may be responsible for the high risk for MS patients to develop depression are unknown.

In this observational study, investigators explore the molecular mechanisms responsible for the impaired regulation of immune cells in relapsing-remitting (RR) MS patients with depression. Investigators will compare the molecular and phenotypical profile of immune cells obtained from RRMS patients with clinical depression (n=50), matched MS patients who do not suffer from depression (n=50) as well as matched healthy controls (n=50) and matched patients with depression but without a comorbid neurological disorder (n=50).

ELIGIBILITY:
Inclusion Criteria:

* Relapsing remitting MS by McDonald Criteria (for RRMS and RRMS+MDD groups).
* Currently meeting diagnostic criteria for Major Depressive Disorder (for MDD and RRMS+MDD groups)
* Age 18-55.
* On stable treatment regime, either untreated or on disease modifying therapy (DMT) for > 6 months

Exclusion Criteria:

* Secondary-progressive or primary progressive MS.
* Substance abuse for more than 6 months.
* Pregnancy
* Use of steroids or vaccination or infections in the previous 3 months.
* Signs of serious psychiatric pathology other than depression including schizophrenia, bipolar disorder or developmental and learning disorders including disorders on the autism spectrum
* Antidepressant medication.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients will be recruited at neurological outpatient clinics and neurologcial clinics of the Charité and neurologists' medical practices.
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Beck Depression Inventory - II | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Friedemann Paul, Prof. Dr., Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité - Universitätsmedizin Berlin, Berlin, Germany

REFERENCES:
- [Background] Dorr J, Ohlraun S, Skarabis H, Paul F. Efficacy of vitamin D supplementation in multiple sclerosis (EVIDIMS Trial): study protocol for a randomized controlled trial. Trials. 2012 Feb 8;13:15. doi: 10.1186/1745-6215-13-15. PMID 22316314
- See also: Related Info — http://dx.doi.org/10.1186/1745-6215-13-15